CLINICAL TRIAL: NCT00257036
Title: A Multicenter, Active-Controlled, Randomized Study to Evaluate the Safety and Efficacy of Levofloxacin Versus Ciprofloxacin HCl in the Treatment of Mild to Moderate Skin and Skin Structure Infections in Adults
Brief Title: A Study of the Safety and Effectiveness of Oral Levofloxacin Compared With Oral Ciprofloxacin in the Treatment of Adults With Mild to Moderate Infections of the Skin and the Supportive Layers Beneath the Skin
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: PriCara, Unit of Ortho-McNeil, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR005476
Record Dates: First submitted 2005-11-18; First posted 2005-11-22 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-01

CONDITIONS: Skin Diseases, Infectious; Cellulitis
Keywords: Infectious skin diseases; skin diseases; bacterial skin diseases; cellulitis; quinolones; levofloxacin
MeSH Terms: conditions — Skin Diseases, Infectious; Cellulitis; Skin Diseases; Skin Diseases, Bacterial | interventions — Levofloxacin

INTERVENTIONS:
Drug: levofloxacin

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of levofloxacin, an antibiotic, compared with ciprofloxacin, another antibiotic, in the treatment of adults with mild to moderate infections of the skin and the supportive layers beneath the skin.

DETAILED DESCRIPTION:
Levofloxacin is an antibacterial agent used for the treatment of many types of infections in adults. This is a randomized, open-label, parallel group, multicenter study to determine the safety and effectiveness of levofloxacin (500 mg by mouth once daily for 7-10 days) compared with another frequently used antibiotic, ciprofloxacin (500 mg by mouth every 12 hours for 7 -10 days), in adults with mild to moderate infections of the skin and the supportive layers beneath the skin. The study consists of 3 visits: one visit [pre-therapy] for screening and enrollment, and two visits to assess safety and effectiveness (one visit [on-therapy] on Days 3 - 5 of the study and one visit [post-therapy] 2 - 7 days after the last dose of the study drug). The total duration of patient participation in the study is approximately 2 weeks. The primary assessments of effectiveness include the clinical response to treatment (defined at post-therapy as cured, improved or failed) and the microbiological response at post-therapy (the rate of eradication of the disease-causing bacteria, determined by patient and by type of bacteria). Safety evaluations (incidence of adverse events, physical examination, physical examination of the skin, and laboratory tests) are performed throughout the study. The study hypothesis is that treatment with levofloxacin is at least as effective and as well tolerated as treatment with ciprofloxacin in patients with mild to moderate infections of the skin and the supportive layers beneath the skin. Levofloxacin 500 mg by mouth once daily, or ciprofloxacin 500 mg by mouth every 12 hours. The duration of treatment is 7 to 10 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mild to moderate infection of the skin and/or the supportive layers beneath the skin, as indicated by pain at the site of the infection, redness, drainage, swelling, or other relevant clinical signs
* tissue sample available from the area of the skin affected by the bacteria
* able to take medication by mouth

Exclusion Criteria:

* Patients with a condition requiring treatment with antibiotics by injection into a vein, a muscle, or beneath the skin
* having a severe infection
* previous allergic or serious adverse reactions to similar antibiotics
* taken antibiotics internally within 48 hours of the start of the study with resulting improvement
* require a second antibiotic taken internally or need an antibiotic applied directly to the site of the infection in addition to the study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 431 (Actual)
Dates: Start 1991-07; Study Completion 1993-02 (Actual)

PRIMARY OUTCOMES:
Clinical response rate (defined as cured, improved or failed) 2 - 7 days after the last dose of the study drug; rate of elimination of disease-causing bacteria (by patient, and by type of bacteria); incidence of adverse events.

SECONDARY OUTCOMES:
Change in physical examination and in laboratory tests after treatment with the study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A study of the safety and effectiveness of oral levofloxacin compared with oral ciprofloxacin in the treatment of adults with mild to moderate infections of the skin and the supportive layers beneath the skin — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=651&filename=CR005476_CSR.pdf